CLINICAL TRIAL: NCT01341093
Title: Educational Program With Telephone Follow-up for Patients After Percutaneous Coronary Intervention: Randomized Controlled Trial
Brief Title: Education Program for Cardiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rejane Kiyomi Furuya, Ph.D, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010/19761-3
Record Dates: First submitted 2011-04-15; First posted 2011-04-25 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Percutaneous Coronary Intervention; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- usual care (Active Comparator)
  Interventions: Behavioral: Usual care
- educational program+telephone follow up (Experimental)
  Interventions: Behavioral: educational program+telephone follow up

INTERVENTIONS:
Behavioral: educational program+telephone follow up — Patients will participate in the educational program with telephone follow-up, the education program will initiate in preoperative period and will continue for six months.
  Arms: educational program+telephone follow up
Behavioral: Usual care — Patients will receive orientations about the surgery and the rehabilitation by health professionals, especially in the discharge. And will have return for evaluation scheduled by health professionals.
  Arms: usual care

SUMMARY:
The purpose of this study is to elaborate an educative program that includes telephone follow-up and assess its impact on the perceived health status of patients submitted to percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or more) of both sexes
* Being submitted to the first coronary artery bypass graft surgery between April 2011 and July 2012
* Having a properly functioning residential phone line

Exclusion Criteria:

* No cognitive condition to participate (assessed through the Mini-Mental State Examination - MMSE)

  * Illiterate participants who did not reach the minimum score 13 on the MMSE
  * Participants with one to seven years of education who did not reach the minimum score 18 on the MMSE
  * Participants with eight or more years of education who did not reach the minimum of 26 points on the MMSE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
change from baseline in perceived health status at six months | baseline and six months
  The questionnaire "Medical Outcomes Survey 36 - Item Short-Form" developed by Ware and Sherboune (1992) will be used to collect the data at baseline and at six months.

SECONDARY OUTCOMES:
change from baseline in treatment adherence at six months | baseline and six months
  The questionnaire "Medida de adesão ao tratamento (MAT)" developed by Delgado and Lima (2001) will be used to collect the data related to the pharmacological adherence at baseline and at six months.
change from baseline in self-efficacy at six months | baseline and six months
  The questionnaire "General Self-Efficacy Scale" developed by Schwarzer and Jerusalem (1995) will be used to collect the data at baseline and at six months.
change from baseline in anxiety and depression at six months | baseline and six months
  The questionnaire "Hospital Anxiety and Depression Scale (HADS)" developed by Zigmond and Snaith (1983) will be used to collect the data at baseline and at six months.

CONTACTS AND LOCATIONS:
Overall Officials: Rejane K. Furuya, PhDCandidate, Principal Investigator — University of São Paulo at Ribeirão Preto College of Nursing; Lidia A. Rossi, PhD, Study Chair — University of São Paulo at Ribeirão Preto College of Nursing
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Furuya RK, Arantes EC, Dessotte CA, Ciol MA, Hoffman JM, Schmidt A, Dantas RA, Rossi LA. A randomized controlled trial of an educational programme to improve self-care in Brazilian patients following percutaneous coronary intervention. J Adv Nurs. 2015 Apr;71(4):895-908. doi: 10.1111/jan.12568. Epub 2014 Nov 17. PMID 25400127